CLINICAL TRIAL: NCT02974439
Title: An Open-Label Randomized, Single-Dose, 2-way Crossover Bioequivalence Study of Amlodipine and Norvasc Under Fasting Condition Sand Under Non-fasting(FED) Conditions in Chinese Healthy Volunteers
Brief Title: Bioequivalence Study of Amlodipine and Norvasc Under Fasting and FED Conditions in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haini Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HN-LD
Record Dates: First submitted 2016-11-17; First posted 2016-11-28 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LANDI-Amlodipine Besylate Tablet 5mg (Experimental): During the study session, healthy subjects will be administered a single dose of LANDI-AmlodipineTablet 5mg under fasting and FED conditions.
  Interventions: Drug: LANDI-Amlodipine Besylate Tablet 5mg
- Norvasc Tablets 5mg (Active Comparator): During the study session, healthy subjects will be administered a single dose of Norvasc Tablets 5mg under fasting and FED conditions.
  Interventions: Drug: Norvasc Tablets 5mg

INTERVENTIONS:
Drug: LANDI-Amlodipine Besylate Tablet 5mg — LANDI-Amlodipine Besylate Tablet 5mg is a generic product manufactured by YangTZE River Pharmaceutical Group Shanghai Haini Pharmaceutical Co., Ltd.
  Other Names: Amlodipine Tablet 5mg
  Arms: LANDI-Amlodipine Besylate Tablet 5mg
Drug: Norvasc Tablets 5mg — Norvasc Tablet 5mg will be used as a comparator drug for the BE study.
  Other Names: Amlodipine Tablet 5mg
  Arms: Norvasc Tablets 5mg

SUMMARY:
This study evaluates the pharmacokinetics and bioequivalence of Amlodipine Besylate Tablets 5 mg versus Norvasc 5 mg tablets administered as 5 mg tablet in healthy volunteers with a washout period of 14 days

DETAILED DESCRIPTION:
The study design is an Open-Label Randomized, Single-Dose, 2-way Crossover Bioequivalence Study with a washout period of 14 days. During each session, the subjects will be administered a single dose of 5mg amlodipine (one LANDI-Amlodipine Tablet 5mg or one Norvasc Tablet 5mg) under fasting and FED conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers of 18-40 years old, male or female.
2. Body mass index (BMI) ranges from 19.0 to 25.0 kg/m2, body weight ≥ 50 kg for male and 45 kg for female.
3. No history of heart, liver, kidney, gastrointestinal tract diseases, nervous system, neural abnormities or metabolic abnormalities; No preparation allergies, serious infection or injury, etc.
4. Medically healthy subjects with clinically normal laboratory profiles and ECGs.
5. Subjects must agree to take effective contraceptive methods to prevent pregnancy from the start of screening until 3 months of last dose administration
6. Subjects are fully informed and voluntarily consent to participate in this study.

Exclusion Criteria:

1. History of allergy or hypersensitivity to amlodipine
2. Significant history of neurological, cardiovascular, digestive, respiratory, urinary, hematological, dysmetabolism or other diseases (such as psychosis) which is unfavorable to the study
3. History of postural hypotension
4. Blood donation or lost more than 400mL blood within 3 months prior to the study
5. Use of medications within 2 weeks before the study
6. Volunteer in any other clinical drug study within 3 months prior to this study
7. Drug abuse or alcohol abuse (220ml beer /day or >5 times in 2 hours)
8. Smoker (>10 cigarettes/day)
9. A positive result in hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, a syphilis test, or an human immunodeficiency virus (HIV) test
10. Abnormal chest X-ray results with clinical significance
11. Women of childbearing potential, pregnant and lactating women.
12. Other unfavorable factors diagnosed by investigators.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Peak Plasma Concentration (Cmax) | 144 hours

SECONDARY OUTCOMES:
Bioequivalence based on Area under the plasma concentration versus time curves (AUC) | 144 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yanmei Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Haini Pharmaceutical Co., Ltd., Shanghai, China

IPD SHARING:
Plan to Share IPD: No